CLINICAL TRIAL: NCT02736253
Title: Determining of Independent Risk Factors for Three Critical Stages of the Diabetic Foot Infections Without Using the Well-known Classification Systems: Osteomyelitis, Amputation and Major Amputation
Brief Title: Risk Factors for Three Critical Stages of the Diabetic Foot Infections
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Serhat Uysal, specialist medical doctor Serhat UYSAL, Ege University
Other Study IDs: 13-1.1/8
Record Dates: First submitted 2016-04-01; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Foot; Osteomyelitis
Keywords: foot amputation; Osteomyelitis; Diabetic Foot
MeSH Terms: conditions — Diabetic Foot; Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study, it was aimed to evaluate the independent risk factors for osteomyelitis, amputation and major amputation of the diabetic foot infection in the forward direction without using standard scoring procedures.

DETAILED DESCRIPTION:
In this study, it was aimed to evaluate the independent risk factors for osteomyelitis, amputation and major amputation of the diabetic foot infection in the forward direction without using standard scoring procedures. Patients who were applied to Diabetic Foot Council of our setting with diabetic foot infections between 2012 and 2014 were included in the study. Patients were followed prospectively and ethical approval was obtained from research ethics committee of our setting. An informed consent form was provided by each patient. Diabetic foot infection was decided as local infection involving only the skin and the subcutaneous tissue or infection involving symptoms and signs more than this criterion. Properties and variables of the cases were recorded during the admission process with total 57 different situations. The related characteristics were followed until the end of the treatment. Osteomyelitis, amputation and factors affecting to have major amputation on the cases were investigated. In the first step, data normality tests were performed with a simple data analysis and univariate analysis was applied in the second stage to which meaningful. At the last stage, major amputation, amputation and osteomyelitis were analyzed with stepwise multiple logistic analysis (SLA) model. Logistic regression was subject as significant data were saved as the independent risk factor. The Odds ratio and 95% CI were calculated from the beta coefficients of the variables with significant p value. P < 0.05 was used for significance at all tests.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in research (An informed consent form was provided by each patient),
* Patient with infected diabetic foot,
* The lack of mental retardation or mental disorders

Exclusion Criteria:

* The patient refused to participate in the study,
* Age < 18 years.
* Patient's opinion or participation in another clinical trial
* The patient has previously been recruited to the study.
* Another rapidly progressive or terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were applied to Diabetic Foot Council of Ege University with diabetic foot infections between 2012 and 2014 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically definite Osteomyelitis | within the first 45 days after admission (hospitalization) (plus or minus 10 days)
  Number of cases with osteomyelitis as assessed with using at least two of criteria below:
  X-ray graphic imaging, magnetic resonance imaging, bone tissue microbiological culture bone pathological biopsy
  Follow-up of patients was completed, after the wound healed. The healing was defined as the complete and uniform skin formation at the wound.
The cases applied amputation(minor or major) and The cases applied major amputation | within the first 3 months after admission
  Transfemoral, transtibial, knee disarticulation, and hipdisarticulation amputations were decided as MAJOR AMPUTATION.
  Other amputation types(more than disarticulation) of lower extremity and major amputations decided as AMPUTATION

SECONDARY OUTCOMES:
To Decide Independent Risk factors for osteomyelitis in patients with Diabetic Foot Infections | within the first 5±2 days after admission
  Data of the cases were recorded during the admission process with total 58 different situations including the demographic data such as age, gender, type of diabetes and the wound characteristics such as length and width of the wound, the laboratory results such as the number of leukocyte, neutrophil percentage and CRP, monitoring results such as osteomyelitis and arterial occlusion, congestive heart failure, comorbid diseases such as cataracts, tissue culture results, results of microbiological examination, Charcot joints or deformity such as claw-foot.
  For determining of data recieved from area of the wound, HD(at least 1900x1080 pixel) images were recorded.
  MDR, XDR, PDR enteric gram-negative microorganisms. MRSA, MRCNS, VRE, ESBL-producer determination factor of any microorganism was adopted as the reproduction of "resistant microorganisms"(1)(2). Fungal growth was recorded also in tissue culture.
To Decide Independent Risk factors for AMPUTATION and - for MAJOR AMPUTATION. | within the first 3 months after admission
  Descriptions were similar with ''Independent Risk factors for osteomyelitis'' But: Osteomyelitis was added to the list(s) for both MAJOR AMPUTATION and AMPUTATION For MAJOR AMPUTATION: AMPUTATION was removed from the list. For AMPUTATION : MAJOR AMPUTATION was removed from the list.

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Uysal, MD, Principal Investigator — Department of Infectious Diseases and Clinical Microbiology, Ege University, Izmir, Turkey; Bilgin Arda, Prof. Dr., Study Director — Department of Infectious Diseases and Clinical Microbiology, Ege University, Izmir, Turkey; Meltem Işıkgöz Taşbakan, Prof. Dr., Study Chair — Department of Infectious Diseases and Clinical Microbiology, Ege University, Izmir, Turkey; Sevki Cetinkalp, Prof. Dr., Study Director — Department of Endocrinology and Metabolism, Ege University, Izmir, Turkey; Ilgin Yildirim Simsir, MD, Study Chair — Department of Endocrinology and Metabolism, Ege University, Izmir, Turkey; Murat Ozturk, MD, Study Chair — Department of Orthopedics and Traumatology, Ege University Medical Faculty, Izmir, Turkey; Ayse Uysal, MD, Study Chair — Department of Internal Medicine, Ege University Medical Faculty, Izmir, Turkey; Ilgen Ertam, Prof.Dr., Study Chair — Department of Dermatology, Ege University Medical Faculty, Izmir, Turkey
Locations (1):
- Ege University Faculty of Medicine, Diabetic Foot Council, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Magiorakos AP, Srinivasan A, Carey RB, Carmeli Y, Falagas ME, Giske CG, Harbarth S, Hindler JF, Kahlmeter G, Olsson-Liljequist B, Paterson DL, Rice LB, Stelling J, Struelens MJ, Vatopoulos A, Weber JT, Monnet DL. Multidrug-resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. Clin Microbiol Infect. 2012 Mar;18(3):268-81. doi: 10.1111/j.1469-0691.2011.03570.x. Epub 2011 Jul 27. PMID 21793988
- [Background] Baio PV, Mota HF, Freitas AD, Gomes DL, Ramos JN, Sant'Anna LO, Souza MC, Camello TC, Hirata Junior R, Vieira VV, Mattos-Guaraldi AL. Clonal multidrug-resistant Corynebacterium striatum within a nosocomial environment, Rio de Janeiro, Brazil. Mem Inst Oswaldo Cruz. 2013 Feb;108(1):23-9. doi: 10.1590/s0074-02762013000100004. PMID 23440110